CLINICAL TRIAL: NCT01868893
Title: An Expanded Access, Open-Label Study of Obinutuzumab (GA101) Plus Chlorambucil in Patients With Previously Untreated Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28979
Record Dates: First submitted 2013-05-29; First posted 2013-06-05 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; Chlorambucil

ARMS (1):
- Obinutuzumab + Chlorambucil (Experimental): Obinutuzumab was administered intravenously for 6 cycles (28-day cycles) as: 100 mg on Day 1, 900 mg on Day 2, and 1000 mg on Days 8 and 15 for Cycle 1; and 1000 mg on Day 1 of Cycles 2 to 6. Chlorambucil was administered orally at a dose of 0.5 mg/kg body weight on Days 1 and 15 for Cycles 1 through 6 (28-day cycles).
  Interventions: Drug: Obinutuzumab; Drug: Chlorambucil

INTERVENTIONS:
Drug: Obinutuzumab
  Other Names: RO 5072759, GA101
Drug: Chlorambucil

SUMMARY:
This is a multicenter, open-label, single-arm, expanded access treatment study designed to provide obinutuzumab to patients with previously untreated Chronic Lymphocytic Leukemia (CLL) in combination with chlorambucil and to evaluate the safety and efficacy of obinutuzumab administered in combination with chlorambucil. This study will enroll patients with previously untreated CD20-positive CLL requiring treatment according to the IWCLL guidelines (Hallek et al 2008), as assessed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CD20-positive CLL (per IWCLL guidelines, Hallek et al 2008)
* Previously untreated CLL requiring treatment according to the IWCLL guidelines (Hallek et al 2008), as assessed by the investigator
* Adequate baseline bone marrow function unless it due to underlying CLL disease No previous treatment for CLL by chemotherapy, radiotherapy, or immunotherapy
* Patients who are not appropriate to receive more intensive chemotherapy in the judgment of the investigator
* Life expectancy of > 6 months

Exclusion Criteria:

* Treatment with any other investigational agent or participation in another clinical trial within 28 days prior to the start of Cycle 1
* Transformation of CLL to aggressive B-cell malignancy History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Known hypersensitivity to chlorambucil or any of its excipients
* History of other malignancy that could affect compliance with the protocol or interpretation of results Known active bacterial, viral, fungal, mycobacterial, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (related to the completion of the course of antibiotics) within 4 weeks before the start of Cycle 1
* Major surgery (within 4 weeks prior to the start of Cycle 1), other than for diagnosis
* Known infection with human immunodeficiency virus (HIV) or Human T-Cell Leukemia Virus 1 (HTLV-1) seropositive status
* Positive hepatitis serology
* Women who are pregnant or lactating
* Fertile men or women of childbearing potential unless 1) surgically sterile or 2) using an adequate measure of contraception such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly
* Effective contraception is required while receiving obinutuzumab. For women, effective contraception is required to continue for >= 12 months after the last dose of obinutuzumab. For men, effective contraception is required to continue for 6 months after the last dose of chlorambucil treatment.
* Vaccination with a live vaccine a minimum of 28 days prior to the start of Cycle 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (19):
- United States (19):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Highlands Oncology Group, Rogers, Arkansas
  - University of California San Diego, La Jolla, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - Cancer Center of Central Conn., Southington, Connecticut
  - Peachtree Hematology & Oncology Consultants, Pc, Atlanta, Georgia
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Kootenai Cancer Center, Coeur d'Alene, Idaho
  - Illinois Cancer Care, P.C. - Galesburg, Galesburg, Illinois
  - Joliet Oncology Hematology Associates, Ltd., Joliet, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Center for Cancer Care, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - San Juan Oncology Associates, Farmington, New Mexico
  - Mark H. Zangmeister Center, Columbus, Ohio
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Northwest Medical Specialties, Tacoma, Washington
  - Vince Lombardi Cancer Clinic Pharmacy, Green Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants were enrolled at 7 study sites in the United States (U.S) between 21 August 2013 and 22 January 2014.
Pre-assignment Details: Of 20 participants, one patient withdrew from the study due to neutropenia and did not receive any study drug.
Period: Overall Study
Arm/Group | Obinutuzumab + Chlorambucil
Started | 20
Completed | 0
Not Completed | 20
Not completed — Adverse Event | 2
Not completed — Commercial availability of study drug | 17
Not completed — Neutropenia | 1

BASELINE CHARACTERISTICS:
Population: Safety population which included all enrolled patients who received at least one dose of study drug (obinutuzumab).
Arm/Group | Obinutuzumab + Chlorambucil
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Obinutuzumab and Chlorambucil in the Study
Description: Number of participants who received obinutuzumab and chlorambucil in the study are presented in the below table.
Time Frame: Cycles 1 to 6 (28-day cycles)
Population: Intent-to-Treat population: It included all enrolled participants in the study.
Measure: Number; unit: participants
Groups:
- Obinutuzumab: Obinutuzumab was administered intravenously for 6 cycles (28-day cycles) as: 100 mg on Day 1, 900 mg on Day 2, and 1000 mg on Days 8 and 15 for Cycle 1; and 1000 mg on Day 1 of Cycles 2 to 6.
- Chlorambucil: Chlorambucil was administered orally at a dose of 0.5 mg/kg body weight on Days 1 and 15 for Cycles 1 through 6.
Arm/Group | Obinutuzumab | Chlorambucil
Number analyzed (Participants) | 20 | 20
participants | 19 | 19

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), AEs of Grade 3 and Above Severity, AEs of Special Interest (AESI), AEs Leading to Obinutuzumab Discontinuation or Dose Delays, Serious Adverse Events (SAEs), and Death
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0 was used for grading the AEs. According to NCI CTCAE, Grade 3 = severe or medically significant but not immediately life threatening; Grade 4 = life-threatening consequences, urgent intervention indicated, and Grade 5 = death. AESIs included all tumor lysis syndrome, serious infections, serious infusion-related reactions (IRR), and hepatitis B reactivation. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to 28 days after the last dose of study drug (up to 7 months from Day 1)
Population: Safety Population: It included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Obinutuzumab + Chlorambucil
Number analyzed (Participants) | 19
participants
  Any AEs | 19
  Any AEs of Grade 3 and more severity | 10
  AEs leading to obinutuzumab discont. or delay | 8
  AESI | 1
  Any SAEs | 2
  Death | 0

3. Secondary Outcome: Number of Participants With Objective Response
Description: Objective response is defined as either complete response [CR], complete response with incomplete recovery [CRi], or partial response [PR] as determined by the treating physician's standard practice at the end of treatment or premature discontinuation from study per the International Workshop on Chronic Lymphocytic Leukemia Criteria (iwCLL criteria). Patients who have not achieved a CR or a PR, and who have not exhibited progressive disease, will be considered to have stable disease (which is equivalent to a nonresponse).
Time Frame: Up to end of treatment or premature discontinuation from study (up to 7 months from Day 1)
Population: Efficacy evaluable population: It included participants who received at least one dose of study drug and had measurable disease at baseline and at least one post-baseline tumor assessment or who died within 28 days after the last dose of the study drug
Measure: Number; unit: participants
Arm/Group | Obinutuzumab + Chlorambucil
Number analyzed (Participants) | 6
participants | 4

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last dose of study drug (up to 7 months from Day 1)
Description: SAEs and other AEs were collected in the safety population, which was defined as all enrolled participants who received at least one dose of study drug.
Arm/Group | Obinutuzumab + Chlorambucil
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + Chlorambucil (N=19)
Anaemia (Blood and lymphatic system disorders) | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Eesophageal ulcers (Gastrointestinal disorders) | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + Chlorambucil (N=19)
Neutropenia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Visual impairment (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Haematochezia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chills (General disorders) | 2
Fatigue (General disorders) | 2
Oedema peripheral (General disorders) | 2
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 12
Fall (Injury, poisoning and procedural complications) | 1
Lymphocyte count decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 3
Glomerular filtration rate decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Weight decreased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 6
Confusional state (Psychiatric disorders) | 1
Bladder pain (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Embolism (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.